CLINICAL TRIAL: NCT06997770
Title: Association Between Grade (B/C)of Stage III and Stage IV Periodontitis and High Sensitivity C Reactive Protein Levels in Serum and Oral Rinse Sample :A Cross Sectional Study
Brief Title: Association Between Grade(B/C)of Stage III and IV Periodontitis and High Sensitivity C Reactive Protein Level in Serum and Oral Rinse Sample
Status: Not yet recruiting | Type: Observational
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: Neha Sahjlan PeriodonticsPGIDS
Record Dates: First submitted 2025-05-12; First posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: hsCRP
Keywords: periodontits

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- generalized periodontitis STAGE III/IV , Grade B: 29 systemically healthy individuals With stage III /IV and grade B
- generalized periodontitis STAGE III/IV , Grade C: 29 systemically healthy individuals With stage III /IV and grade C
- Periodontally healthy individuals: 29 systemically and periodontally healthy individuals

SUMMARY:
According to 2017 World Workshop of Periodontology , the level of high sensitivity C reactive protein has been assumed to increase according to the grade of periodontitis, however, specific evidence regarding this is lacking at present. Hence, measuring high sensitivity C reactive protein in serum and oral rinse samples in systemically healthy individuals with periodontitis could be potentially useful in gaining insight on the systemic burden of periodontal disease.

DETAILED DESCRIPTION:
According to 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions , the level of high sensitivity c reactive protein has been assumed to increase according to the grade of periodontitis, however, specific evidence regarding this is lacking at present. Moreover, no information is currently available regarding the feasibility of detecting high sensitivity in oral rinse samples, which are relatively easy to collect and store, as compared to more commonly investigated oral fluids like saliva and gingival crevicular fluid Previous literature reports that saliva and gingival crevicular fluid levels of high sensitivity C reactive protein correlate with serum high sensitivity C reactive protein levels, therefore, there is a possibility that high sensitivity C reactive protein in oral rinse samples might also be correlated with serum high sensitivity C reactive protein levels. Measuring high sensitivity C reactive protein in serum and oral rinse samples in systemically healthy individuals with periodontitis could be potentially useful in providing easily accessible information about the systemic burden of periodontal inflammation as well as regarding detection of subclinical systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients in the age group of (18-50 years)
* Presence of ≥ 20 natural teeth
* Ability and willingness to give written informed consent
* Patients belonging to 3 groups -periodontally healthy, stage III and stage IV grade B periodontitis, and stage III and stage IV grade C periodontitis .

Exclusion Criteria:

* • Patients with chronic inflammatory disease such as nephrotic syndrome, chronic renal failure, significant cardiovascular disease, established type 1 or type 2 diabetes mellitus, or active cancer within the past 5 years

  * Smokers and alcoholics
  * Pregnant females
  * Presence of xerostomia
  * Patients undergoing radiotherapy
  * Having received professional periodontal treatment within the previous 6 months
  * Having received antibiotic medication 3 months prior to study
  * Periapical pathology or other oral inflammatory conditions
  * Cognitive disability (interfering with ability to give sample)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 1. Group 1: comprising of periodontally healthy individuals.
  2. Group 2: comprising of individuals, diagnosed with stage III and stage IV grade B periodontitis (according to WWP 2017 classification periodontal disease )
  3. Group 3: comprising of participants, diagnosed with stage III and IV grade C periodontitis,
Sampling Method: Probability Sample
Enrollment: 87 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-08-25 (Estimated)

PRIMARY OUTCOMES:
Evaluation of hscrp level in oral rinse samples and serum in 3 groups of systemically healthy individuals | 12-14 months
  Evaluation of hsCRP level in oral rinse samples and serum in 3 groups of systemically healthy individuals (periodontally healthy, stage III and stage IV grade B generalized periodontitis, stage III and stage IV grade C generalized periodontitis)

SECONDARY OUTCOMES:
Correlation of Probing pocket depth (PPD)and Clinical attachment level (CAL) with level of hsCRP in oral rinse and serum samples. | 12-14 months
  Correlation of Probing pocket depth (PPD) with level of hsCRP in oral rinse and serum samples.
  Correlation of Clinical attachment level (CAL) with level of hsCRP in oral rinse and serum samples.
Correlation of Bleeding on probing (BOP%) | 12-14 months
  Correlation of Bleeding on probing (BOP%) with level of hsCRP in oral rinse and serum samples.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Aditi Sangwan, MDS, Principal Investigator — PGIDS ,ROHTAK
Locations (1):
- PGIDS, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No